Preoperative Gabapentin versus Bisoprolol for hemodynamic and surgical field optimization during Endoscopic Sinus Surgery: randomized controlled trial

By

- 1. Abeer M. Elnakera<sup>1</sup>
- 2. Maram H. Wagdy<sup>2</sup>
- 3. Aymen A. Abd-Elgelyl<sup>2</sup>
- 4. Mohamed W. EL-Anwar<sup>3</sup>

NCT03850093

Document Date: December 15, 2016

## **Statistical methods:-**

Continuous parametric data were presented as mean and standard deviation (SD) and compared using one way ANOVA (F) followed by pos-hoc analysis for intergroup comparison and repeated measures of ANOVA was used for intragroup comparison. Quantitative non-parametric data were presented as median and range and compared using kruskal Wallis test. Qualitative data were presented as number and percentage and compared using Chi-square test ( $X^2$ ). P value < 0.05 was considered significant and all statistical methods were 2 tailed. Statistical analysis was performed in SPSS version 24